CLINICAL TRIAL: NCT03544671
Title: Effect of Vitamin D3 Supplementation Over 25-hydroxivitamin D (25-OH-D) Status in Children From 12-30 Months of Age: Randomized Clinical Trial
Brief Title: Effect of Vitamin D3 Supplementation in Children From 12 to 30 Months of Age.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Mario Flores-Aldana, Mario Flores-Aldana, MD, PhD Nutrition Surveillance, Director, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114-7000
Record Dates: First submitted 2018-05-17; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Vitamin D Deficiency; 25-Hydroxyvitamin D3 Deficiency, Selective
Keywords: Vitamin D; Nutritional deficiencies; Miconutrients; Children; Mexico
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin D Hydroxylation-Deficient Rickets, Type 1B; Malnutrition | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel, controlled trial was conducted in children from 12 to 30 months of age who received four supplements. Four treatments groups were assign randomly to children: One group received 400 IU/d, the second group received 800IU/d of vitamin D2 and the third one 1,000IU/d of colecalciferol D3. The fourth group-control-group- received a multy vitamin supplementation containing: iron, vitamin A, C, and E, folic acid, niacin and vitamins B1, B2, B6 y B12.Children were enrolled from 14-day-care centers which are part of a national government program Secretaria de Desarrollo Social "SEDESOL" , which main objective is to support working mothers and those who intend to work and do not have access to a health service.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Moses Oakford method was used by an independent researcher to randomly assign each child to 1 of 3 groups to receive the administration of the three supplments. A computer was used to generate the random numbers (STATA v.13). Groups were stratified by age from 12- 18 months, from 19- 24 months and form 25- 30 months of age. Each block group was assigned 73 children.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 400 IU/d vitamin D2 (Experimental): Children received 1mililiter (dosage applicator) containing 400 IU of vitamin D2 per day. This suplement also contained: iron, vitamin A, C, and E, folic acid, niacin and vitamins B1, B2, B6 y B12. Vitamin D2, dosage form (1 mililiter), frequency (daily) and duration 16 weeks
  Interventions: Dietary Supplement: Vitamin D
- 800 IU7d vitmin D2 (Experimental): Children received 2 mililiter (dosage applicator) containing 800 IU of vitamin D2 per day. This suplement also contained: iron, vitamin A, C, and E, folic acid, niacin and vitamins B1, B2, B6 y B12. Vitamin D2, dosage form (1 mililiter), frequency (daily) and duration 16 weeks
  Interventions: Dietary Supplement: Vitamin D
- 1000 IU vitamina D3 (Experimental): Children received 1drop (dosage applicator) containing 1000 IU of vitamin D3 per day. dosage form (1 drop), frequency (daily) and duration 16 weeks
  Interventions: Dietary Supplement: Vitamin D
- Multiple vitamin (Placebo Comparator): Children received 1 mililiter of a supplement with multiple vitamins (dosage applicator) frequency (daily) and duration 16 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D

SUMMARY:
Background Vitamin D (VD) is essential for calcium absorption, bone health and growth in children. In a national representative sample authors found mean serum concentration of 25-Hydroxi-Vitamin-D (25-OH-D) of 59 nmol/L, in children < 5 y of age. Prevalence deficiency of VD under 50 nmol/L was 33%, which means that 3 million preschool- age children have VD deficiency in Mexico. Additionally, less than 3% of the children use supplements with VD.

Objective To assess the effect of 400UI, 800IU of vitamin D2 and 1000IU of vitamin D3-colecalciferol- over 25-Hidroxi Vitamin D (25-OH-D) status and a multiple vitamin supplementation per day as a control group in children from 12-30 months of age in Cuernavaca, Morelos in a 4 month period.

Methods Randomized double blind parallel clinical trial, with vitamin D3 (colecalciferol) supplementation in 220 children from 12 - 30 months who attend day care centers.

Three supplementations will be given to children: 400IU and 800IU of vitamin D2, the third group 1000IU of D3-colecalciferol- and the control group will receive a multi vitamin supplementation. The duration of the intervention will be 16 weeks. Blood measurements would be taken at baseline, and at 16 weeks.

This study compares the efficacy of three dose of VD in children from 12-30 months of age, over the nutritional status of 25 hydroxivitamin D (25-OH-D). This intervention is of importance to establish supplementation strategies to prevent VD deficiency in Mexico.

Keywords: Vitamin D, nutritional deficiencies, micronutrients, children, México.

DETAILED DESCRIPTION:
2. Objective. To assess the effect of 400UI, 800IU of vitamin D2 and 1000IU of vitamin D3-colecalciferol- over 25-Hidroxi Vitamin D (25-OH-D) status and a multiple vitamin supplementation per day as a control group in children from 12-30 months of age in Cuernavaca, Morelos in a 4 month period.

3. Hypothesis Supplementation with 1,000 IU/d of vitamin D3-colecalciferol will have a greater effect on 25-OH-D concentrations compared to a dose of 400 IU and 800IU per day of vitamin D2 and will be more effective to decrease vitamin D deficiency in children from 12-30 months of age 4. Methods. 4.1 Study design. Factorial randomized double blind, parallel, controlled clinical trial with administration of a supplement containing 400IU or 800 IU of D2 or 1,000 IU of vitamin D3 -colecalciferol- and a multiple vitamin supplementation per day as a control group during a 4 month period.

Participants: A total of 220 children, both sexes, from 12-30 month of age will be studied (55 per treatment group).

Intervention period: 4 months Project duration: 18 months Place: Day Care centers(SEDESOL) in Cuernavaca, Morelos 4.2. Treatment: The Moses Oakford method will be used to assign the treatment. The scheme to randomize the sample will be by stratification and in blocks using a list of random numbers generated by a computer (STATA13). Stratification will be by age groups 12-18 months, 19-24 months and 25-30 months. Treatment will be assigned randomly to each supplement group. One group will receive 400IU of vitamin D2, the second group will receive 800 IU of D2, the third group will receive 1000IU of D3-colecalciferol- and the control group will receive a multi vitamin supplementation, that contains iron, vitamin A, C. E folic acid, niacin, and vitamins B1, B2, B6 y B12 The duration of the intervention will be 16 weeks.

4.3. Study Population- Children between 12 and 30 months of age, both sexes, which attend day care centers that are part of a national government program which main objective is to support working mothers and those who intend to work and do not have access to a health service. The program also includes single parents in charge of their family. Sample will be by convenience until sample is completed. Day care will be selected by convenience, (Principal interested in participating in the research project). A reunion will be made with authorities from SEDESOL and with the principals of the day care centers. The study objective, methodology and the importance of the project will be explained. After the meeting, a list of the day care centers who wish to participate will be made. A meeting with the parents will be assigned in order to explain the purpose, importance, objective and methods of the project.

Inclusion Criteria. Children- from 12-30 months of age, both sexes who attend SEDESOL day care centers in Cuernavaca, and whose parents agree to participated and sign the informed consent.

Exclusion Criteria. Chronic disease, anemia (Hb<9.0), does not want to participate, receiving vitamin D supplementation or other supplement in the last 6 months.

4.4. Sample size and statistical power. Up to date, efficacy studies on vitamin D supplementation in preschool-age children are scarce. Three studies were considered: The sample size of these studies have been around 100-150 children in total.

The first study supplemented preschool-age children with 400IU of vitamin D for 4 months, having found a positive difference on the supplemented group of 23 nmol/L of 25-OH-D in relation with the placebo group. The second study was carried out with infants, the aim of the study was to test the efficacy, dose response of various international units of vitamin D: 400, 800, 1,200 and 1,600 per day with a follow up of 12 months. The increase in serum levels of 25-OH-D were: 18, 42, 74 y 120 nmol/L, respectively. On the other hand, other study supplemented children between 2 weeks and 3 months of age with various doses of vitamin D daily for 3 months: 400, 1,200 ó 1,600 IU/d. The increases observed in serum levels of 25-OH-D in this study were: de 14, 37.5 y 66.5 nmol/L, respectively.

Considering these studies, and the serum levels of 25-OH-D observed in our study in the same population during 2012(41-50 nmol/L), it is expected to observe an increase around 20 nmol/L in children receiving 400 IU/d and de 40 nmol/L in children receiving 1,000 IU/d of VD.

The size and power of the sample was calculated considering a basal level of serum 25-OH-D of 41 a 50 nmol/L with an increase of 20-40 nmol/L with a S.D of 20 a 40 nmol/L. As a result, a sample size of 100 children per group were obtained. With this sample a mean difference of 10 nmol/L can be obtained with a power of 80% α<0.05-two tails- 4.5. Variables. Outcome variables. Measurements will be taken at base line and at 16 weeks: serum 25-OH-D, parathyroid hormone (PTH) and hemoglobin.

Other variables. Anthropometry: Anthropometric measurements such as: weight, height/length, head circumference and mid upper arm will be taken. Measurements will be taken by trained and standardized personnel using standard technics according to protocols. Measurements will be taken at baseline and at 16wk. Weight, height/length and circumferences will be transformed to Z scores by using the Anthro WHO program.

Diet: Dietary information will be obtained by a food frequency questionnaire (FFQ) and a 24-h recall. Both dietary questionnaires will be administered by trained personnel to the mother/care taker. Dates will be set with mothers in these two momentums to obtain dietary information. Dietary information will be taken at baseline and at 16wks.

Morbidity: Morbidity data will be collected daily at each day care center by trained personnel. A checklist will be used to record symptoms of diarrhea and acute respiratory infections. Mothers or caretakers will be asked to recall any symptoms.

Sociodemographic Characteristics: Information about the participant's household's characteristics, the education level and parents occupation will be obtained by interviewing of the mother. An indicator of household conditions will be calculated by principal component analysis.

Infant Development:

A screening test will be applied to assess and identified children at risk. This test is called in spanish "Prueba Evaluacion Desarrollo Infantil" (EDI).

4.6 Statistical Analysis. The effect of the intervention over the final serum concentrations of 25-OH-D will be evaluated through a t test for median differences. If the variables do not have a normal distribution, will be transformed. If important differences are found at the beginning of the study between treatment groups, a multiple linear regression will be made to control for confounding variables.

4.7. Study Stages and Data Collection. 4.7.1 Recruitment Recruitment and follow-up of children will be made at the day-care centers (SEDESOL) in Cuernavaca, Morelos. A date will be established at each day care center to explain to mothers the study objective and procedures: anthropometric, biochemical, diet, socioeconomic questionnaire, randomization and treatment. A consent form will be read to each parent and signed if accept to participate. Doubts will be cleared at the meeting with parents.

4.7.2 Baseline Anthropometric measurements will be taken: Weight, length/height, head and mid upper arm circumferences. During the first visit capillary blood samples will be taken in situ to measure hemoglobin concentrations (Hb) by a spectrophotometer Hemocue®. According to selection criteria if a child has <9.0g/dl, the child will be referred to the nearest health center. A vein blood sample (5mL) will be taken to determine serum concentrations of 25-OH-D y PTH. The sample will be obtained by a Pediatrician Nurse with experience. A sosciodemographic questionnaire will be applied to obtain information on household, education, marital status and income. In this first visit, children will be randomly assigned to the treatment. All interviews and measurements will be taken by trained and standardized personnel.

4.7.3 Intervention: Treatment will be administered according to randomization: 400IU/d, 800IU/d, 1000 IU/d and a multivitamin. Two standardized and trained personnel will be present each day at each day care center. With a list of the names of the participants in hand each child will be called to receive the assigned treatment. Every day at 7:00 a.m. children will receive the treatment.

4.7.4 Adverse effects: The maximum dose -1,000 IU/d- it's under the upper level UL, according to the recommendations of the Institute of Medicine (IOM) for children between 12 and 36 months of age. By definition the "Upper Level" it's considered a safe intake by the IOM expert comity therefore, adverse effects associated with 1,000 IU7d will not be observed for prolonged periods at this age group.

4.7.5 Toxicity Monitoring: Every day at 7:30 a.m. a trained nutritional student will be gathering morbidity information and adverse effects. The adverse effects associated with excessive intake of vitamin D are: dehydration, nausea, vomiting, conscious alterations and high calcium excretion. If symptoms were to appear, a medical pediatrician will monitor and follow the child. High calcium excretion it is only observed in severe intoxication with vitamin D.

If adverse effects were to appear in the study population, the researchers responsible of the study will stop the study and report adverse effects.

4.7.6 Committee experts on adverse effects: The committee experts will be held by Dr. Patricia Clark and Dr. María Dolores Ramirez. Assessment of adverse effects will be held at the National Institute of Public Health in Cuernavaca, Morelos, Mexico.

4.7.7 Final Assessment A meeting will be held with each mother at each day care center to obtain information on child´s diet. A 24 Hour recall and a Frequency Food Questionnaire will be applied to the mother. The last assessment will be at 16 weeks. Anthropometric measurements will be taken: Weight, length/height, head and mid upper arm circumferences.

Blood Samples Capillary blood samples will be obtained by finger prick and measured in a Portable Photometer Hemocue. Venous blood samples (5ml) will be drawn from antecubital vein at baseline at 16wks. Samples will be obtained by a trained Pediatrician Nurse who has previews experience working with children.

5. Ethical considerations: Written Informed consent will be obtained and signed by both parents. The study protocol is approved by the Ethics, Research and Biosecurity Committee of the National Institute of Public Health.

ELIGIBILITY:
Inclusion Criteria:

Children form 12-30 months of who attend the day care centers Children whose parents accepted their child to participate and sign the informed consent

Exclusion Criteria:

* Children receiving multiple micronutrient supplementation/ other vitamin D suplement
* Children whose parents did not accept to participate
* Children with capillary hemoglobin concentration <9.0 g/dL at baseline

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-06-18 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Chanche in 400UI,of vitamin D2 over 25-Hidroxi Vitamin D | Measurements were taken at baseline, and at 16 weeks
  nmol/L
Chanche in 800UI,of vitamin D2 over 25-Hidroxi Vitamin D | Measurements were taken at baseline, and at 16 weeks
  nmol/L
Change in 1000 of vitamin D3 over 25-Hidroxi Vitamin D | Measurements were taken at baseline, and at 16 weeks
  nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Mario Flores, PhD, Principal Investigator — National Institute of Public Health, Mexico
Locations (1):
- Marta Rivera Pasquel, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No